CLINICAL TRIAL: NCT04065867
Title: SMART Family-Link Project: Using Information and Communication Technology to Improve Family Interventions and Promote Family Well-being in Hong Kong
Brief Title: Use ICT to Promote Family Well-being in Hong Kong
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: The Hong Kong Jockey Club Charities Trust (Other)
Responsible Party: Sponsor
Other Study IDs: UW 19-489
Record Dates: First submitted 2019-08-20; First posted 2019-08-22 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Family Relations
Keywords: Family

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: ICT activities — Family interventions using ICT to promote family communication, sharing happiness with family members, and well-being in the community.

SUMMARY:
In the past few decades, Information and Communications Technology (ICT) have rapidly developed as effective, and probably the most cost-effective tools to connect most aspects of family lives. Alongside the growth in popularity of ICTs and its role in promoting family well-being, there is also an increasing appreciation that ICTs such as internet-enabled devices and web-based applications can offer many advantages compared to traditional face-to-face approaches when delivering behaviour change programmes.

To gain more understanding of the potential new avenues of using ICT in programme implementation, The Hong Kong Jockey Club Charities Trust has initiated the Jockey Club SMART Family-Link Project in collaboration with The University of Hong Kong (HKU) and non-governmental organizations (NGOs). This project aimed at helping 26 NGO-operated Integrated Family Service Centres and Integrated Service Centres (Centres), making effective use of information and communications technology (ICT) and data analytics, to enhance the quality and efficiency of their family service. The present study aims to supplement the existing services and interventions delivered by the FRU, FSU and FCU, a series of brief ICT-based family interventions that promote family communication, cohesion, support and well-being and improve the efficiency and effectiveness of ICT-based interventions.

DETAILED DESCRIPTION:
Information and communications technology (ICT) as a global trend The last few decades have seen a dramatic rise in the use of information and communications technology (ICT) and Internet access. According to the World Bank, 1.33 per cent of individuals in the world were using the Internet in 1996; in 2006, this figure rose to 17.58 %; by 2016, 45.91 % of individuals were using the Internet. Concurrently, there has been a dramatic rise in the number of mobile cellular subscriptions across the globe in the last two decades.

In line with the global trend, Hong Kong had 18.25 million mobile service subscribers in 2016. The Hong Kong Family and Health Information Trends Survey (FHinTs) under the Jockey Club FAMILY Project was conducted to monitor opinions and behaviours regarding family health, information use, and health communications. Our results showed that ICT platforms such as online websites, social media, and instant messages are widely used in Hong Kong. In FHinTs 2016 survey, 82.6% of the respondents had smartphones, and 48.8% had tablets. Similar findings from the Nielsen Media Index 2017 year-end report showed that 97% of all internet users in Hong Kong were using smartphones to access the internet. The amount of time spent online each day was 3.2 hours and 94% of people aged 12 to 64 were using the internet.

The role of ICT in enhancing family well-being in Hong Kong With the increasing use of ICT, family information can be easily accessed. According to the findings from FHinTs 2016, ICT was increasingly used as a method of family information seeking: 66.7% of respondents sought family information from online websites, compared with 53.6% in 2009. About 30.9% sought family information from social media such as Facebook, and 22.8% sought family information from instant messaging platforms such as WhatApp. Family information such as recreation (46.6%), family heath (22.9%) and elderly-related topics (17.9%) were most commonly sought. Also, family information seeking was associated with higher levels of family health, happiness, harmony, and overall family well-being. The associations were observed regardless of the type of sharing methods, such as face-to-face sharing or sharing via ICT means.

ICT in family interventions Alongside the growth in popularity of ICTs and its role in promoting family well-being, there is also a growing appreciation that ICTs such as internet-enabled devices and web-based applications can offer many advantages compared to traditional face-to-face approaches when delivering behaviour change programmes.

One of the biggest challenges of face-to-face programmes is diminishing reach and impact due to barriers to accessibility, cost-efficiency, flexibility to adapt to individuals, and structured intervention integrity . Using ICTs can address these barriers and may thus contribute to improving reach. ICT also helps facilitate access to interventions from a large variety of settings at all times, bringing the intervention to participants at times convenient to them and diminishing the influence of the situational constraints on intervention participation rates. The rise of ICT has created promising and potential new avenues and demand for implementing interventions related to mental health and parenting.

Family services in Hong Kong In light of the review on family services in Hong Kong in 2000, pilot projects on the Integrated Family Service Centre (IFSC) service mode were conducted in 2002. Having received positive feedback from the community on the pilot projects, 61 IFSCs were established in 2004 to provide public-funded family services in Hong Kong. These IFSCs comprise three important components, including the family resource unit (FRU), family support unit (FSU), and family counselling unit (FCU) to provide preventive, supportive, and remedial services respectively. They are operated by the Social Welfare Department and subvented non-governmental organizations to support and strengthen individuals and families, particularly single parents, new arrivals, ethnic minorities, and deprived families receiving Comprehensive Social Security Assistance (CSSA), in the community.

Society is always changing, and so do the community and families. In order to meet the changing needs of the community and families, a Review on the Implementation of the IFSC service mode was carried out in 2008 and completed in 2010 to evaluate the effectiveness of the IFSC service mode. The Review report "Building Effective Family Services: Review on the Implementation of the IFSC Service Mode" stated that the IFSC service mode is an appropriate service mode for public-funded family services in Hong Kong. However, the Review also identified factors hindering the delivery of IFSC services. These hindering factors are namely poor accessibility of some IFSCs, heavy workload, and stigmatization. With the use of ICT, these hindering factors can be overcome, thus improving the IFSC service mode.

Jockey Club SMART Family-Link Project Family well-being is the cornerstone of a harmonious society, and early support for families in need will avert crisis. The Hong Kong Jockey Club Charities Trust has funded to a four-year (2018-2021) "Jockey Club SMART Family-Link Project" to advance the use of Information and Communications Technology ("ICT") in family services. Interventions leveraging ICT (i-Action) is one of the project components, which leverage ICT to help social workers offer ICT-based interventions in their work to add on their face-to-face interventions. ICT tools and mobile apps will be designed and interactive games will be provided to engage children and young family service users through e-platforms. Social workers will also be able to connect with service users between face-to-face sessions using these e-platforms.

Importance of this study The present study aims to supplement the existing services and interventions delivered by the FRU, FSU and FCU, a series of brief ICT-based family interventions that promote family communication, cohesion, support and well-being and improve the efficiency and effectiveness of ICT-based interventions.

This protocol is to seek approval from Institutional Review Board (IRB) to collect data from the participants in the family services for in-depth analysis, and to write up scientific papers based on the findings generated from this project.

ELIGIBILITY:
Inclusion Criteria:

* Family service users
* Chinese-speaking
* Aged 18 years and above
* Able to complete the questionnaire

Exclusion Criteria:

* Subjects who fail to meet the inclusion criteria

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Social service users
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2019-09-09 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Satisfaction to the family services | Immediately after the activities
  Outcome-based questions will be used to assess the level of satisfaction toward the general performance of the community activities. The score for each question ranges from 1 to 5. The higher score indicates the higher satisfaction.

SECONDARY OUTCOMES:
Family communication | Baseline, immediately after activities and 1 month
  Outcome based question will be used to assess the communication with family members. The score for each question ranges from 0 to 10. The higher score indicates the better family communication.
ICT use in sharing | Baseline and immediately after activities
  Outcome based questions will be used to assess the attitude and practice on sharing happiness with family members and friends. The score for each question ranges from 0 to 10. The higher score indicates the better outcome performance
Family relationship | Baseline and 1 month
  Outcome based question will be used to assess the relationship with family members. The score for each question ranges from 0 to 10. The higher score indicates the better family relationship.
Family happiness | Baseline and 1 month
  Outcome based question will be used to assess the family happiness.The score for question ranges from 0 to 10. The higher score indicates the better in family happiness
Parenting | Baseline, immediately after activities and 1 month
  Outcome based question will be used to assess the parenting.The score for question ranges from 0 to 10. The higher score indicates the better parenting.
Family support and care | Baseline, immediately after activities and 1 month
  Outcome based question will be used to assess the family support and care.The score for question ranges from 0 to 10. The higher score indicates the more family support and care.
Resilience | Baseline, immediately after activities and 1 month
  Outcome based question will be used to assess the resilience.The score for question ranges from 0 to 10. The higher score indicates the higher resilience.
Healthy living habits | Baseline and 1 month
  Outcome based question will be used to assess the healthy living.The score for question ranges from 0 to 10. The higher score indicates the more healthy living.
Social connectedness | Baseline, immediately after activities and 1 month
  Outcome based question will be used to assess the social connectedness.The score for question ranges from 0 to 10. The higher score indicates the more social connectedness.
Personal happiness | Baseline and 1 month
  Outcome based question will be used to assess the personal happiness.The score for question ranges from 0 to 10. The higher score indicates the better in personal happiness

CONTACTS AND LOCATIONS:
Overall Officials: Tai-hing Lam, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Background] Breitenstein SM, Gross D, Christophersen R. Digital delivery methods of parenting training interventions: a systematic review. Worldviews Evid Based Nurs. 2014 Jun;11(3):168-76. doi: 10.1111/wvn.12040. Epub 2014 May 19. PMID 24842341
- [Background] Enebrink P, Hogstrom J, Forster M, Ghaderi A. Internet-based parent management training: a randomized controlled study. Behav Res Ther. 2012 Apr;50(4):240-9. doi: 10.1016/j.brat.2012.01.006. Epub 2012 Jan 30. PMID 22398153
- [Background] Gross D, Johnson T, Ridge A, Garvey C, Julion W, Treysman AB, Breitenstein S, Fogg L. Cost-effectiveness of childcare discounts on parent participation in preventive parent training in low-income communities. J Prim Prev. 2011 Dec;32(5-6):283-98. doi: 10.1007/s10935-011-0255-7. PMID 22134677
- [Background] Kingston D, Janes-Kelley S, Tyrrell J, Clark L, Hamza D, Holmes P, Parkes C, Moyo N, McDonald S, Austin MP. An integrated web-based mental health intervention of assessment-referral-care to reduce stress, anxiety, and depression in hospitalized pregnant women with medically high-risk pregnancies: a feasibility study protocol of hospital-based implementation. JMIR Res Protoc. 2015 Jan 16;4(1):e9. doi: 10.2196/resprot.4037. PMID 25595167
- [Background] Bert SC, Farris JR, Borkowski JG. Parent training: implementation strategies for adventures in parenting. J Prim Prev. 2008 May;29(3):243-61. doi: 10.1007/s10935-008-0135-y. PMID 18446440
- [Background] Treisman GJ, Jayaram G, Margolis RL, Pearlson GD, Schmidt CW, Mihelish GL, Kennedy A, Howson A, Rasulnia M, Misiuta IE. Perspectives on the Use of eHealth in the Management of Patients With Schizophrenia. J Nerv Ment Dis. 2016 Aug;204(8):620-9. doi: 10.1097/NMD.0000000000000471. PMID 26828911
- [Background] Proudfoot J. The future is in our hands: the role of mobile phones in the prevention and management of mental disorders. Aust N Z J Psychiatry. 2013 Feb;47(2):111-3. doi: 10.1177/0004867412471441. No abstract available. PMID 23382507
- See also: Hong Kong Communications Authority, 2016. Telecommunications — http://www.gov.hk/en/about/abouthk/factsheets/docs/telecommunications.pdf
- See also: The World Bank, 2016. Internet users (per 100 people) — http://data.worldbank.org/indicator/IT.NET.USER.P2?end=2014&start=1990